CLINICAL TRIAL: NCT00915096
Title: High Tumor Burden Follicular Lymphoma: Impact of [18F]-FDG Positron Emission Tomography (PET) in the Assessment of Treatment Response
Brief Title: Positron Emission Tomography (PET)-Scan in the Evaluation of High Tumor Burden Follicular Lymphoma
Status: Completed | Type: Observational
Sponsor: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Other Study IDs: PET-FOL
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma, Follicular
Keywords: Follicular Lymphoma; PET; GELA
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Burden tissue sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High Tumor Burden Follicular Lymphoma

SUMMARY:
The purpose of the study is to assess in a prospective series of patients with high tumor burden follicular lymphoma treated with R-CHOP, the predictive value of [18F]-FDG PET performed over (after 4 treatments), and at the end of the first-line treatment on progression-free survival at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant non-Hodgkin follicular lymphoma (histologic grade 1 to 3 in the WHO classification), histologically confirmed,
* Patients who have not previously been treated for this disease,
* Introducing one of the criteria for high tumor burden,
* Patients aged over 18 and under 80 years,
* Patients whose ECOG condition is ≤ 2,
* Patients whose haematological functions are adequate within 28 days preceding the treatment (Hemoglobin ≥8,0g/dl; Neutrophils ≥1,5e-9/L, Platelets ≥100e-9/L),
* Patient had the PET examination less than a month before the start of chemotherapy.

Exclusion Criteria:

* Patients with lymphoma who have already transformed or been treated for this disease,
* Patients whose lymphoma is stage 3b,
* Patients with impaired central nervous system,
* Patients regularly taking corticosteroids during the 4 weeks preceding the treatment (unless the dose administered is equivalent to ≤20 mg/day prednisone).
* Patients who have undergone major surgery during the 28 days preceding the inclusion,
* Patients with low kidney and/or liver function,
* Patients with HIV + or had an infection with HBV or HCV less than 4 weeks. Patients with hepatitis B serology is positive unless the sign is related to vaccination,
* Patients whose life expectancy ≤ 6 months,
* Patients sensitive or allergic to murine products,
* Patients who participated in another clinical trial during the 30 days preceding the recording,
* Patients with other medical problems or psychological succeptibles interfere with the study,
* Patients under adult supervision.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High Tumor Burden Follicular Lymphoma patients
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2007-09-18 (Actual); Primary Completion 2011-05-10 (Actual); Study Completion 2013-02-08 (Actual)

PRIMARY OUTCOMES:
Predictive value of PET on progression-free survival | 2 years

SECONDARY OUTCOMES:
Comparison of PET results to treatment response (Cheson criteria) | 30 weeks
Correlation of PET data with FLIPI index score | Baseline
Comparison of changes in lymph node volumes measured by CT to changing of FDG fixation | 30 weeks
Correlation of PET data with histopathological data (including the use of immunohistochemical markers) | Baseline
Evaluation of the sensitivity of PET in the detection of the involvement of hematopoietic marrow | Baseline
Comparison of conventional criteria for evaluating the response to the criteria "revised" by the international workshop criteria | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michel MEIGNAN, Prof, Principal Investigator — Lymphoma Study Association; Jehan DUPUIS, MD, Principal Investigator — Lymphoma Study Association
Locations (22):
- France (21):
  - CHU - Besançon, Besançon
  - CHU Avicenne, Bobigny
  - Centre Bergognié, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - Clinique Victor Hugo, Le Mans
  - Centre Hospitalier - Lens, Lens
  - CHRU Lille, Lille
  - CHU - Limoges, Limoges
  - Centre Paoli-Calmettes, Marseille
  - CHU - Nantes, Nantes
  - Hôpital Necker, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Saint-Louis, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - CHU Purpan, Toulouse
  - Hôpital Bretonneau, Tours
  - CHU Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Ospedale Cuneo, Cuneo, Italy

REFERENCES:
- [Derived] Dupuis J, Berriolo-Riedinger A, Julian A, Brice P, Tychyj-Pinel C, Tilly H, Mounier N, Gallamini A, Feugier P, Soubeyran P, Colombat P, Laurent G, Berenger N, Casasnovas RO, Vera P, Paone G, Xerri L, Salles G, Haioun C, Meignan M. Impact of [(18)F]fluorodeoxyglucose positron emission tomography response evaluation in patients with high-tumor burden follicular lymphoma treated with immunochemotherapy: a prospective study from the Groupe d'Etudes des Lymphomes de l'Adulte and GOELAMS. J Clin Oncol. 2012 Dec 10;30(35):4317-22. doi: 10.1200/JCO.2012.43.0934. Epub 2012 Oct 29. PMID 23109699
- See also: GELA — http://www.gela.org